CLINICAL TRIAL: NCT02285153
Title: Does Acetylsalicylic Acid Reduce the Mortality of Patients Admitted to an Intensive Care Unit
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment of planned number of Subjects was not feasible.
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Bernd Jilma, Ao. Univ.-Prof. Dr. Bernd Jilma, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASA-MORT; 2012-002235-29 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2014-11-06 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Critical Illness
Keywords: acetylsalicylic acid; intensive care unit; mortality; Post mortem examination; bleeding
MeSH Terms: conditions — Critical Illness; Hemorrhage | interventions — acetylsalicylic acid lysinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetylsalicylic acid lysinate (Experimental): 100mg Acetylsalicylic Acid
  Interventions: Drug: Acetylsalicylic acid lysinate
- 0.9% sodium-chloride solution (Placebo Comparator): 0.9% sodium-chloride solution
  Interventions: Drug: 0.9% sodium-chloride solution

INTERVENTIONS:
Drug: Acetylsalicylic acid lysinate — 100mg intravenously administered Acetylsalicylic Acid lysinate per day
  Arms: Acetylsalicylic acid lysinate
Drug: 0.9% sodium-chloride solution — Placebo, intravenously administered, daily
  Arms: 0.9% sodium-chloride solution

SUMMARY:
Platelets play a central part not just in homeostasis and thrombosis as the primary effector cells, but they are also key cells in the regulation of the immunological response to various stressors. After activation, platelets release their granules which store different inflammatory mediators that induce coagulation, recruit further platelets, activate complement, attract neutrophils and leukocytes and regulate the vascular tone. Platelets activated by systemic inflammation and infection, may also contribute to the development of multiple organ failure. Thus, inhibition of platelet activation may have beneficial effects on critically ill patients.

the investigators hypothesize that acetylsalicylic acid reduces the mortality of medical intensive care unit patients. In a retrospective study acetylsalicylic acid use was associated with a substantial reduction in a medical intensive care unit population (Winning et al., 2010).

The investigators will conduct a randomized, double-blind study including 460 patients (2x230), who will be randomized to receive 100mg acetylsalicylic acid(daily, intravenous) or a placebo (0,9% sodium-choride solution) to assess whether acetylsalicylic acid reduces the mortality of medical intensive care unit patients.

Main outcome criteria will be 28/90day-mortality. Furthermore the investigators will assess whether acetylsalicylic acid reduces the risk of suffering thromboembolic complications.

Post-mortem examinations will be conducted in all patients who die in the course of the study.

Furthermore we will assess bleeding rates, intensive care unit mortality and pharmacokinetic and pharmacodynamic properties of acetylsalicylic acid in the intensive care unit population.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to an intensive care unit
* >18 years of age

Exclusion Criteria:

* known allergy of intolerance to acetylsalicylic acid
* recent surgery or planned surgery
* active bleeding
* known coagulation disorders
* discretion of the physician
* terminal illness (anticipated life expectancy <3months; e.g. due to cancer)
* platelet count <20 000
* recent ulcera
* recent gastrointestinal bleeding
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11-15 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, Ao. Univ.-Prof. Dr. med, Principal Investigator — Medical University of Vienna, Department of Clinical Pharmacology
Locations (1):
- General Hospital, Vienna, Austria

REFERENCES:
- [Background] Winning J, Neumann J, Kohl M, Claus RA, Reinhart K, Bauer M, Losche W. Antiplatelet drugs and outcome in mixed admissions to an intensive care unit. Crit Care Med. 2010 Jan;38(1):32-7. doi: 10.1097/CCM.0b013e3181b4275c. PMID 19770746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetylsalicylic Acid Lysinate | 0.9% Sodium-chloride Solution
Started | 7 | 8
Completed | 6 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetylsalicylic Acid Lysinate | 0.9% Sodium-chloride Solution | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 2 | 4 | 6
Age, Continuous [Median (Standard Deviation); unit: years] | 61 (15) | 63 (10) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 6 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 7 | 8 | 15
Simplified Acute Physiology Score III [Median (Standard Deviation); unit: score on a scale] — The Simplified Acute Physiology Score III is a commonly used disease severity score specifically designed for critically ill patients. It was calculated on the day of admission The score may range from 0 to 217 points. The score includes information on conditions that led to ICU admission, underlying diseases, ventilation, catecholamine use, laboratory data Higher scores predicted mortality, while lower scores were associated with survival.
  score on a scale | 64 (19) | 63 (13) | 64 (15)

OUTCOME MEASURES:

1. Primary Outcome: 28-day Mortality
Description: Standard outcome measure of investigational intensive care unit trials.
Time Frame: 28-days
Population: modified Intention to treat population (all patients who received at least a single dose of acetylsalicylic acid)
Measure: Number; unit: participants
Arm/Group | Acetylsalicylic Acid Lysinate | 0.9% Sodium-chloride Solution
Number analyzed (Participants) | 7 | 8
participants | 1 | 1
Statistical Analysis 1: Comparison: Acetylsalicylic Acid Lysinate vs 0.9% Sodium-chloride Solution; Test type: Superiority; p = 0.57, Chi-squared — Due to the low number of participants, the results of the statistical tests must be interpreted with caution!; Cox Proportional Hazard = 0.434, 95% CI 2-sided [0.039 to 4.792], Standard Error of Mean 1.225

2. Secondary Outcome: Intensive Care Unit Mortality
Description: Mortality of patients during their intensive care unit stay, 90 day mortality, potentially longer
Time Frame: up to 90 days after inclusion
Measure: Number; unit: participants
Arm/Group | Acetylsalicylic Acid Lysinate | 0.9% Sodium-chloride Solution
Number analyzed (Participants) | 7 | 8
participants | 2 | 1
Statistical Analysis 1: Comparison: Acetylsalicylic Acid Lysinate vs 0.9% Sodium-chloride Solution; Test type: Superiority; p = 0.057, Chi-squared

3. Secondary Outcome: Number of Patients Who Developed a Thrombotic or Embolic Complications During the Trial
Description: clinically relevant thromboembolic events assessed by standard care, potentially longer
Time Frame: average 28 days
Measure: Number; unit: participants
Arm/Group | Acetylsalicylic Acid Lysinate | 0.9% Sodium-chloride Solution
Number analyzed (Participants) | 7 | 8
participants | 0 | 1
Statistical Analysis 1: Comparison: Acetylsalicylic Acid Lysinate vs 0.9% Sodium-chloride Solution; Test type: Superiority; p = 1, Chi-squared

4. Secondary Outcome: Bleeding Incidences
Description: all bleeding incidence during the intensive care unit stay will be recorded. major bleeding criteria are taken from the Thrombolysis in myocardial infarction study (TIMI-Triton-38), potentially longer
Time Frame: average 28days
Measure: Number; unit: counts
Arm/Group | Acetylsalicylic Acid Lysinate | 0.9% Sodium-chloride Solution
Number analyzed (Participants) | 7 | 8
counts | 1 | 0
Statistical Analysis 1: Comparison: Acetylsalicylic Acid Lysinate vs 0.9% Sodium-chloride Solution; Test type: Superiority; p = 0.467, Chi-squared

ADVERSE EVENTS:
Time Frame: Duration of the Trial: Inclusion until ICU discharge, up to 365 days
Description: mortality was the primary endpoint. Therefore death was treated as an endpoint rather than a serious adverse event.
Arm/Group | Acetylsalicylic Acid Lysinate | 0.9% Sodium-chloride Solution
All-Cause Mortality (participants affected / at risk) | 2/7 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/8
Other Adverse Events (participants affected / at risk) | 4/7 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetylsalicylic Acid Lysinate (N=7) | 0.9% Sodium-chloride Solution (N=8)
Asystolia (Cardiac disorders) | 1 (1) | 0 (0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
hypoxic brain damage (Nervous system disorders) | 0 (0) | 1 (1)
Colon Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Catheter infection (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetylsalicylic Acid Lysinate (N=7) | 0.9% Sodium-chloride Solution (N=8)
Bleeding (Vascular disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Delirium (Nervous system disorders) | 2 (2) | 1 (1)
Nausea (General disorders) | 0 (0) | 1 (1)
Obstipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
catheter infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes Virus Infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study had to be terminated because of a poor recruitment rate. Thus, all results need to be interpreted with great caution. Patients were critically ill. Hence, the occurrence of adverse events should be interpreted accordingly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02285153/Prot_SAP_000.pdf